CLINICAL TRIAL: NCT05409768
Title: Comparison of Short Axis Out of Plane Method and Anteroposterior Short Axis in Plane Method in Ultrasound-guided Central Venous Catheterizations
Brief Title: Comparison of Two Approach in Ultrasound Guided Central Venous Catheterizations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ilker Ital, Assistant Professor Doctor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AIBU-TF-AR-II-001
Record Dates: First submitted 2022-05-08; First posted 2022-06-08 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Central Venous Catheterization
Keywords: Ultrasound Guided Short; Central Venous Catheterization; Short Axis in-plane
MeSH Terms: interventions — Aircraft

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Short axis, out of plane approach (Experimental): A linear ultrasound probe will be utilized to place the central catheter into the jugular vein with a short axis out of the plane method
  Interventions: Procedure: Short axis out of plane
- Short axis, anteroposterior in plane approach (Experimental): A linear ultrasound probe will be utilized to place the central catheter into the jugular vein with an anteroposterior short axis in-plane method
  Interventions: Procedure: Anteroposterior short axis in plane

INTERVENTIONS:
Procedure: Short axis out of plane — A standard 20 cm (adult-size) 3-port central catheter will be placed to the indicated patients by using standard Seldinger technique (with the assist of a guide wire) under ultrasound guidance short axis visualisation out of plane approaches.
  Other Names: Ultrasound guided central venous catheterization with short axis out of plane approach
  Arms: Short axis, out of plane approach
Procedure: Anteroposterior short axis in plane — A standard 20 cm (adult-size) 3-port central catheter will be placed to the indicated patients by using standard Seldinger technique (with the assist of a guide wire) under ultrasound guidance anteroposterior short axis visualisation in plane approaches.
  Other Names: Ultrasound guided central venous catheterization with anteroposterior short axis in plane approach
  Arms: Short axis, anteroposterior in plane approach

SUMMARY:
Ultrasound guidance in central venous catheterization has become the standard for clinical practice. Many approaches have been described in ultrasound guided catheterization procedures. The aim of this study is to compare the classical short axis out of plane (SAX-OOP) approach and the new anteroposterior short axis in plane (APSAX-IP approach in central jugular venous catheterization. The study was planned as prospective randomized and controlled. One hundred patients were planned to be included in this study.

Patients will be divided into two groups: Central jugular vein catheterization will be performed with the short axis out of plane group (ultrasound transducer will be positioned classically from medial to lateral in the neck) and anteroposterior short axis in plane group (ultrasound transducer will be positioned laterally from anterior to posterior on the neck). The two groups will be compared in terms of number of puncture attempts, duration of the procedure, ultrasound scan time before the procedure, number of needle redirection, overall success rate, complications, ease of catheterization and ultrasound visibility.

DETAILED DESCRIPTION:
Central venous catheterization is a method frequently used in intensive care patients and patients to be operated. With classical methods, this central venous vascular access procedure in the landmark method can be performed or it can be successfully performed under ultrasound guidance.

Ultrasound-guided central venous catheterization is a safer and recommended approach. During venous catheterization with ultrasound the vein and its neighborhood can be easily visualized and it can be followed while the needle is directed to the target in vein puncture. Undesirable complications (hematoma, pneumothorax, arterial puncture) also decrease with the decrease in the number of punctures under ultrasound guidance. Ultrasound guided central catheterization which facilitates safer and faster procedures constitutes an important area for patient care. With the development of technology and the increase in accessibility it constitutes an important and useful area in the interventions made with ultrasound. The internal jugular vein is a frequently chosen central venous structure.

Many ultrasound-guided imaging and intervention methods have been described for catheterization of the internal jugular vein with the Seldinger method. These are described as longitudinal (long axis), transverse (short axis) and oblique methods for imaging and probe position. The image taken with the position of the needle relative to the ultrasound probe is described as in plane and out of plane.

Each method may have advantages over each other and can be preferred according to the patient's condition and the experience of the practitioner. Successful and safe catheterizations can be performed in the internal jugular vein with the short axis out-of-plane (SAX-OOP) method which is especially used in adults . Short axis out of plane is a successful method that can almost be called a classic that comes to mind first. Compared to other needle imaging methods out of plane tracking of the needle (as a point) seems to be a disadvantage in the user's imaging compared to the in-plane tracking method. Of course, it is easier and faster to capture the short axis when imaging the venous structure as long axis or short axis with ultrasound.

The " Anteroposterior short axis in plane" (APSAX-IP) technique is first reported by Aithal G. et al. in 2019. The use of both short axis and in-plane approaches has been described.The difference of the anteroposterior short axis in plane (APSAX-IP ) technique from the classical short axis out of plane (SAX-OOP) technique is that the location of the ultrasound is lateral to the neck, the needle is about 2-3 cm away from the ultrasound, the entry area from the skin, the needle is advanced subcutaneously in the anteroposterior direction, not medially, and the needle is not as a point in ultrasound that can be viewed longitudinally. It is thought that the APSAX-IP method has advantages such as easier follow-up of the needle, easier monitoring of the progression of the needle without damaging the posterior wall by seeing a large anterior posterior diameter of the vessel. It is stated that the APSAX-IP method will be more ergonomic in patients with short neck anatomy, obese and pediatric patients due to the location of the ultrasound probe. One method may be preferred over the other in patients. Although the definition of the method has been made, it has not been compared with any catheterization method. The aim of our study is to compare the classical SAX-OOP method and the newly defined APSAX-IP method in terms of difficulty, needle puncture time, needle procedure time and complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are planned a central venous catheter placement

Exclusion Criteria:

* Morbid obese patients (body mass index> 40)
* People with severe coagulopathy
* Severe deformity at the neck
* Skin deformity or infection at catheterization site
* Congenital anomalies of central veins
* Emergency operations

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-09-10 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of puncture attempts | From the 1st second through withdrawal of the needle, up to 3 minutes
  Number of needle insertions to the catheterization region for placing a catheter
Cannulation procedural time | During the procedure, starting from the 1st second through placement of the catheter; up to 3 minutes
  Duration of the whole cannulation procedure
Catheterization procedural time | During the procedure, starting from the 1st second through placement of the catheter; up to 3 minutes
  Duration of the whole catheterization procedure
Number of needle redirections | During the whole cannulation procedure
  Redirections of the needle towards the vessel
Success rate | Through catheterizations completion, an average of 4 months
  Correct placement of the catheter over the guidewire after central vein puncture
Success rate at first attempt | Through study completion, an average of 4 months
  Success rate at first attempt of the procedures in each group
Complications | Through study completion, an average of 4 months ]
  Rate of complications that occur during catheterization procedure

SECONDARY OUTCOMES:
Vessel visualization | Throughout the procedure; up to 3 minutes
  Visualization of the vessels in dynamic ultrasound images
Needle visualization | Throughout the procedure; up to 3 minutes
  Visualization of the needle in dynamic ultrasound images
Guide-wire visualization | Throughout the procedure; up to 3 minute
  Visualization of the guide-wire in dynamic ultrasound images
Ease of the catheterization process | Throughout the procedure; up to 3 minutes
  A subjective score assigned by the operator on a scale with a minimum value of 0 and maximum value of 10. Higher scores mean a better outcome
Ultrasound time | Throughout the pre-procedural ultrasonography; up to 10 minutes
  The duration of pre-procedural ultrasound scanning

CONTACTS AND LOCATIONS:
Overall Officials: Ilker Ital, MD, Principal Investigator — Bolu Abant Izzet Baysal University Medical School
Locations (2):
- Turkey (Türkiye) (2):
  - Abant İzzet Baysal Education and Training Hospital, Bolu, Merkez
  - Bolu Abant İzzet Baysal University Faculty of Medicine, Bolu

REFERENCES:
- [Background] Aithal G, Muthuswamy G, Latif Z, Bhaskaran V, Haji Sani HS, Shindhe S, Manap NBA, Vadaje KS, Dato Paduka Buntar WS, Daiwajna RG. An Alternate In-Plane Technique of Ultrasound-Guided Internal Jugular Vein Cannulation. J Emerg Med. 2019 Dec;57(6):852-858. doi: 10.1016/j.jemermed.2019.08.029. Epub 2019 Oct 18. PMID 31635927
- [Background] Ince I, Ari MA, Sulak MM, Aksoy M. [Comparison of transverse short-axis classic and oblique long-axis "Syringe-Free" approaches for internal jugular venous catheterization under ultrasound guidance]. Braz J Anesthesiol. 2018 May-Jun;68(3):260-265. doi: 10.1016/j.bjan.2017.12.002. Epub 2018 Feb 23. PMID 29478705
- [Background] Aydin T, Balaban O, Turgut M, Tokur ME, Musmul A. A Novel Method for Ultrasound-Guided Central Catheter Placement-Supraclavicular Brachiocephalic Vein Catheterization Versus Jugular Catheterization: A Prospective Randomized Study. J Cardiothorac Vasc Anesth. 2022 Apr;36(4):998-1006. doi: 10.1053/j.jvca.2021.06.010. Epub 2021 Jun 12. PMID 34247928
- [Background] Rossi UG, Rigamonti P, Ticha V, Zoffoli E, Giordano A, Gallieni M, Cariati M. Percutaneous ultrasound-guided central venous catheters: the lateral in-plane technique for internal jugular vein access. J Vasc Access. 2014 Jan-Feb;15(1):56-60. doi: 10.5301/jva.5000177. Epub 2013 Oct 7. PMID 24101418
- [Background] Troianos CA, Hartman GS, Glas KE, Skubas NJ, Eberhardt RT, Walker JD, Reeves ST; Councils on Intraoperative Echocardiography and Vascular Ultrasound of the American Society of Echocardiography; Society of Cardiovascular Anesthesiologists. Special articles: guidelines for performing ultrasound guided vascular cannulation: recommendations of the American Society of Echocardiography and the Society Of Cardiovascular Anesthesiologists. Anesth Analg. 2012 Jan;114(1):46-72. doi: 10.1213/ANE.0b013e3182407cd8. Epub 2011 Nov 29. No abstract available. PMID 22127816